CLINICAL TRIAL: NCT06172686
Title: Adaptation of Blood-stage Controlled Human Malaria Infection for Evaluation of Transmission Blocking Malaria Interventions in Malaria Endemic Countries
Brief Title: In-vivo Transmission Model in Semi-immune Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ifakara Health Institute (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Blood-CHMI Trans
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Controlled Human Malaria Infection; Induced Blood Stage Malaria Infection; Malaria Transmission; Malaria Challenge
MeSH Terms: interventions — piperaquine; Doxycycline

STUDY DESIGN:
Intervention Model Description: Two antimalarial drugs will be used to induce gametocytes. The first arm will receive Piperaquine tablets (Piramal Pharma Solutions, India), that will be administered orally. Sub-curative regimen will be given as two tablets of 320mg and 160mg (total of 480mg). The second arm will receive Doxycycline (100mg tablets strength as Doxycycline hyclate) that will also be administered orally. Sub-curative regimen will be given as 1 tablet (100mg) once daily for 7 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1 (Experimental): The first arm will receive Piperaquine tablets , that will be administered orally. Sub-curative regimen will be given as two tablets of 320mg and 160mg (total of 480mg).
  Interventions: Drug: Piperaquine tablets , which will be administered orally as a single dose of 480mg (320mg+160mg).
- Arm 2 (Experimental): The second arm will receive Doxycycline (100mg tablets strength as Doxycycline hyclate) that will also be administered orally. Sub-curative regimen will be given as 1 tablet (100mg) once daily for 7 days.
  Interventions: Drug: Doxycycline (100mg tablets strength as Doxycycline Hyclate) will also be administered orally and will be given as 1 tablet (100mg) Once daily for 7 days.

INTERVENTIONS:
Drug: Piperaquine tablets , which will be administered orally as a single dose of 480mg (320mg+160mg). — The first arm will receive Piperaquine tablets, that will be administered orally. Sub-curative regimen will be given as two tablets of 320mg and 160mg (total of 480mg).
  Arms: Arm1
Drug: Doxycycline (100mg tablets strength as Doxycycline Hyclate) will also be administered orally and will be given as 1 tablet (100mg) Once daily for 7 days. — The second arm will receive Doxycycline (100mg tablets strength as Doxycycline hyclate) that will also be administered orally. Sub-curative regimen will be given as 1 tablet (100mg) once daily for 7 days.
  Arms: Arm 2

SUMMARY:
Controlled human malaria infection (CHMI) has revolutionized the development of malaria vaccines. It involves the administration of either known numbers of sporozoites or infected erythrocytes to healthy human volunteers under a controlled environment. The use of highly sensitive molecular malaria diagnostic methods informs treatment decisions before symptom development and allows the characterization of parasite growth dynamics. Sporozoite CHMI has safely been used in six countries in Africa providing a platform to assess the efficacy of candidate malaria vaccines and study the natural immunity to malaria. Blood stage CHMI involves administration of known number of Artemether Lumefantrine sensitive infected erythrocytes in healthy volunteers, and it is a more sensitive model for modelling parasite growths and study the efficacy of blood-stage malaria vaccines. It has been safely used in Australia and Europe but not in Africa. Adaptation of this model by administration of combination of suboptimal and optimal antimalarial drugs lead to increased gametocytaemia, and infection rates in mosquitoes following standard membrane feeding assay. Such adaptation allows the model to be used to study parasite transmission from human to mosquitoes and evaluate transmission blocking malaria interventions.

There is an urgent need to establish an in vivo model for early-stage clinical evaluation of transmission blocking interventions (TBI) in volunteers living in malaria endemic countries. This would allow rapid and cost-effective way to down-select transmission blocking candidate malaria vaccine and gametocidal antimalarial drugs before larger, more complex, and expensive field efficacy studies are conducted. A study done in naïve individual showed 100% success in establishing a malaria infection using 2800 P. falciparum infected RBCs, while a recent study (manuscript in development) has demonstrated success in establishing infection in Tanzanian semi-immune individuals with low malaria exposure using 1000 P. falciparum infected RBCs. We will use 1000 ALU-sensitive 3D7 P. falciparum infected RBCs to establish an in vivo transmission model for studying Transmission blocking interventions and assess the efficiency of two antimalarial drugs regimens (Piperaquine and doxycycline) to induce high levels of gametocytaemia and mosquito infection rates in healthy African adults. We will also investigate the determinants of successful transmission to mosquitoes including underlying immune responses to both asexual and sexual malaria antigens, asexual parasite dynamics and gametocyte burden, sex ratio of male and female gametocytes, and the relationship between gametocyte density and mosquito infection rate

DETAILED DESCRIPTION:
Adaptation of blood-stage Controlled Human Malaria Infection for evaluation of transmission blocking malaria interventions in malaria endemic countries.

This will be Phase I Randomized open label trial. It will recruit Healthy male adults aged 18-45 years from low malaria endemic area (Bagamoy0) for three months.

BACKGROUND AND RATIONALE Plasmodium falciparum (Pf) malaria remains a disease of public health significance affecting millions across the globe (1). Scaling up of malaria interventions has reduced the malaria burden in several parts of Africa (2-5), but this has not been consistent everywhere, with some areas reporting sustained or even an increase in the burden of malaria (6, 7). Vaccination is one of the most cost-effective public health interventions (8, 9) and would play a critical role in the elimination efforts. There is a significant development in research to identify promising transmission-blocking malaria vaccines, with several candidate vaccines in the pipeline. To down-select the most promising candidates, antibody tests and functional assays that prevent infection of mosquitoes are normally used (10). It is however unclear how well these assays represent the in vivo transmission-blocking efficacy making it difficult to choose which candidate to develop further (11). Before a transmission blocking vaccine (TBV) can be approved, a randomized trial to evaluate the effect on gametocyte carriage and transmission to mosquitoes or Phase 3 trial to demonstrate vaccine impact on the incidence of infection in the target population are required. Both study designs are large and expensive (11). Alternatively, accelerated approval could be sought through surrogate markers of efficacy that would require either analytical or biological, but not clinical validation. However currently there is no known surrogate markers. Therefore, in vivo transmission blocking model for early-stage clinical evaluation of TBV is needed to rapidly down-select promising candidate vaccines before large field trials are conducted. Although such model has been studied in malaria naïve population, it is important to establish this model in target populations to provide relevant results that considers the genetic background and underlying natural immunity.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged 18-45 years and in good health.
* Volunteer has adequate understanding of the procedures of the study and is able and willing (in the investigator's opinion) to comply with all study requirements.
* Participant is willing and able to give informed consent for participation in the trial.
* Participant with low malaria exposure as determined by anti-schizont ELISA
* Literacy in Kiswahili.
* Anti-schizont antibody levels below 50th centile of the most recently available population anti-schizont in Bagamoyo district

Exclusion Criteria:

* Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, gastrointestinal, renal, hepatic, neurological, dermatological (e.g. psoriasis, contact dermatitis etc.), allergy, endocrine, malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results.
* A heightened risk of cardiovascular disease, as determined by: an estimated ten-year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiac events in 1st or 2nd degree relatives <50 years old.
* Body mass index (BMI) of <18 or >30 Kg/m2
* A medical history of functional asplenia
* Female volunteers
* Confirmed parasite positive by PCR a day before challenge i.e., at C-1.
* Screening tests positive for Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV)
* Chronic use (>30 days) of i) immunosuppressive drugs, ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral antihistamines exempted) or expected use of such during the study period
* Any recent (within 30 days) or current systemic therapy with an antibiotic or drug with potential antimalarial activity (chloroquine, doxycycline, tetracycline, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, erythromycin, hydroxychloroquine, etc.) (Allowable time frame for use at the Investigator'sdiscretion).
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.
* Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.
* History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
* Previous participation in any malaria investigational product study (allowable time frame for use at the Investigator's discretion)
* Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
* Being an employee or relative of an employee of Ifakara Health Institute.
* Current participation in another clinical trial or recent participation within 12 weeks of enrolment.
* Prior receipt of an investigational malaria vaccine.
* Previous receipt of malaria sporozoites (PfSPZ) or infected RBC as part of the malaria challenge study.
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
* Confirmed parasite positive by qPCR at screening (can be treated and rescreened if time allows)
* History of epilepsy in the period of five years prior to study onset, even if no longer on medication.
* Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.
* History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
* Known hypersensitivity to or contra-indications (including co-medication) for use of Piperaquine, doxycycline, chloroquine, primaquine, artemether-lumefantrine or history of severe (allergic) reactions to blood transfusion.
* Any other condition or situation that would, in the opinion of the investigator, place the volunteer at an unacceptable risk of injury or render the volunteer unable to meet the requirements of the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-09 (Estimated); Primary Completion 2024-02-13 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Solicited and unsolicited adverse events | Up to day 98 after blood infection challenge.
  Frequency of solicited and unsolicited adverse events.
Magnitude of Adverse Events | Up to day 98 after blood infection challenge.
  Magnitude of Adverse Events both solicitated and Unsolicited

SECONDARY OUTCOMES:
Rate of Mosquito infections (proportion of infected mosquitoes) | 14, 21 and 28 days after infection challenge
  Rate of Mosquito infections (proportion of infected mosquitoes)
Infection burden (Oocysts density in infected mosquitoes) | 14, 21 and 28 days after infection challenge
  Infection burden (Oocysts density in infected mosquitoes)
Number of volunteers in each study arm that show prevalence of gametocytes as defined by quantitative reverse-transcriptase PCR (qRT-PCR) for CCp4 (female) and pfMGET (male) mRNA with a threshold of 5 gametocytes/mL for positivity. | Up to day 28 after blood infection challenge
  Number of volunteers in each study arm that show prevalence of gametocytes as defined by quantitative reverse-transcriptase PCR (qRT-PCR) for CCp4 (female) and pfMGET (male) mRNA with a threshold of 5 gametocytes/mL for positivity.
Time to peak density gametocytes from the time of challenge as measured by qRT-PCR. | Up to day 28 after the blood infection challenge
  Time to peak density gametocytes from the time of challenge as measured by qRT-PCR.
The area under the curve of gametocyte density versus time for both arms of the study | Up to day 28 after the blood infection challenge
  The area under the curve of gametocyte density versus time for both arms of the study
Gametocyte commitment after the blood infection challenge as estimated by dividing the peak gametocyte by the peak of asexual parasites | Up to day 28 after the blood infection challenge
  Gametocyte commitment after the blood infection challenge as estimated by dividing the peak gametocyte by the peak of asexual parasites
Gametocyte Sex-ratio after blood infection challenge as measured by the proportion of male gametocytes versus female gametocytes. | Up to day 28 after the blood infection challenge
  Gametocyte Sex-ratio after blood infection challenge as measured by the proportion of male gametocytes versus female gametocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Ally Olotu, MD,Dphil, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Pwani, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the de-identified data on the parasite dynamics and safety of volunteers who participated in the study. This will be done during publication of the study results.
Supporting Information: Study Protocol
Time Frame: within 12 months after study completion
Access Criteria: Open access

REFERENCES:
- [Background] Aregawi MW, Ali AS, Al-mafazy AW, Molteni F, Katikiti S, Warsame M, Njau RJ, Komatsu R, Korenromp E, Hosseini M, Low-Beer D, Bjorkman A, D'Alessandro U, Coosemans M, Otten M. Reductions in malaria and anaemia case and death burden at hospitals following scale-up of malaria control in Zanzibar, 1999-2008. Malar J. 2011 Feb 18;10:46. doi: 10.1186/1475-2875-10-46. PMID 21332989
- [Background] Ceesay SJ, Casals-Pascual C, Nwakanma DC, Walther M, Gomez-Escobar N, Fulford AJ, Takem EN, Nogaro S, Bojang KA, Corrah T, Jaye MC, Taal MA, Sonko AA, Conway DJ. Continued decline of malaria in The Gambia with implications for elimination. PLoS One. 2010 Aug 18;5(8):e12242. doi: 10.1371/journal.pone.0012242. PMID 20805878
- [Background] Farnert A, Yman V, Homann MV, Wandell G, Mhoja L, Johansson M, Jesaja S, Sandlund J, Tanabe K, Hammar U, Bottai M, Premji ZG, Bjorkman A, Rooth I. Epidemiology of malaria in a village in the Rufiji River Delta, Tanzania: declining transmission over 25 years revealed by different parasitological metrics. Malar J. 2014 Nov 26;13:459. doi: 10.1186/1475-2875-13-459. PMID 25423887
- [Background] Okiro EA, Hay SI, Gikandi PW, Sharif SK, Noor AM, Peshu N, Marsh K, Snow RW. The decline in paediatric malaria admissions on the coast of Kenya. Malar J. 2007 Nov 15;6:151. doi: 10.1186/1475-2875-6-151. PMID 18005422
- [Background] Assele V, Ndoh GE, Nkoghe D, Fandeur T. No evidence of decline in malaria burden from 2006 to 2013 in a rural Province of Gabon: implications for public health policy. BMC Public Health. 2015 Feb 4;15:81. doi: 10.1186/s12889-015-1456-4. PMID 25649228
- [Background] Okiro EA, Bitira D, Mbabazi G, Mpimbaza A, Alegana VA, Talisuna AO, Snow RW. Increasing malaria hospital admissions in Uganda between 1999 and 2009. BMC Med. 2011 Apr 13;9:37. doi: 10.1186/1741-7015-9-37. PMID 21486498
- [Background] Holden JD. Benefits and risks of childhood immunisations in developing countries. Br Med J (Clin Res Ed). 1987 May 23;294(6583):1329-31. doi: 10.1136/bmj.294.6583.1329. PMID 3109642
- [Background] Robertson RL, Foster SO, Hull HF, Williams PJ. Cost-effectiveness of immunization in The Gambia. J Trop Med Hyg. 1985 Oct;88(5):343-51. PMID 3939146
- [Background] Miura K, Swihart BJ, Deng B, Zhou L, Pham TP, Diouf A, Burton T, Fay MP, Long CA. Transmission-blocking activity is determined by transmission-reducing activity and number of control oocysts in Plasmodium falciparum standard membrane-feeding assay. Vaccine. 2016 Jul 29;34(35):4145-4151. doi: 10.1016/j.vaccine.2016.06.066. Epub 2016 Jun 29. PMID 27372156
- See also: World Health O. World malaria report 2019. Geneva: World Health Organization; 2019 2019 — http://www.who.int/publications/i/item/9789241565721